CLINICAL TRIAL: NCT02538991
Title: TVT Versus Bulkamid®-Injections in Treatment of Stress Urinary Incontinence - Patient Satisfaction and Complications of the Treatment
Brief Title: TVT Versus Bulkamid®-Injections in Treatment of Stress Urinary Incontinence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anna-Maija Itkonen, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/13/03/03/2015
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Urinary Stress Incontinence
Keywords: Bulkamid; Tension-Free Vaginal Tape; Women
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

ARMS (2):
- Bulkamid (Experimental)
  Interventions: Device: Bulkamid
- Tension-free Vaginal Tape (Active Comparator)
  Interventions: Device: Tension-free Vaginal Tape

INTERVENTIONS:
Device: Bulkamid — Urethral injections will be performed policlinically under local anesthesia (10 ml lidocain, two injections on both sides of the urethra). The Bulkamid-injections will be transurethral four injections (0.2 - 1ml) in locations "ten, two and five and seven o'clock" within 0.5 to 1 cm from the bladder - urethra junction.
  Additional injections will be avoided and can be injected only if the first injections fail. After the operation the patient urinates to empty the bladder. The PVR is checked after the treatment with ultrasound simultaneously with evaluation of stability of the Bulkamid-injections. The treatment will be photographed as before and after still pictures for later evaluation.
  Arms: Bulkamid
Device: Tension-free Vaginal Tape — TVT will be performed under local anesthesia (70 - 100 ml 0.25% prilocain cum epinephrine) with i.v. pain medication phentanyl two doses and more on request. Operation will be performed with TVT-Exact® kit. Operation can be performed policlinically or in an operation theatre depending on the patient's medical condition. Cystoscopy will be performed after the set of tapes. A cough stress test with 250 to 300 ml bladder fulfillment will show the right tension of the tape. Before the operation a prophylactic antibiotic of Cefuroxime 1.5 g i.v will be given (Dalacin 900 mg i.v in cases of allergy to penicillin). The patient can go home after 2 to 4 hours follow-up, when PVR is under 150 ml. A sick leave of 5 days is recommended.
  Arms: Tension-free Vaginal Tape

SUMMARY:
One out of three adult females suffer from daily urinary incontinence. Two thirds of urinary incontinence is physical activity-related stress urinary incontinence (SUI). If the first-line treatment for SUI, training of pelvic floor muscles, is insufficient, treatment options are suburethral sling operation or transurethral bulking injection. Randomized studies between TVT and Bulkamid® and the knowledge about cost-effectiveness and patient satisfaction is missing.

This prospective randomized study compares TVT and Bulkamid®-injections in treatment of SUI. Main outcome measures are patient satisfaction, complications and effectiveness of the treatment in reducing urinary leakage. Secondary outcome measures are cost-effectiveness, pain during and after treatment and changes in Quality of Life and symptoms.

DETAILED DESCRIPTION:
1. Background

   One out of three adult females suffer from daily urinary incontinence. Two thirds of urinary incontinence is physical activity-related stress urinary incontinence (SUI). If the first-line treatment for SUI, training of pelvic floor muscles, is insufficient, treatment options are suburethral sling operation or transurethral bulking injection.

   Tension-free Vaginal Tape (TVT) is considered the gold standard for the treatment of SUI1. TVT operation is an effective treatment with efficacy as high as 90%. TVT performed by an experienced operator carries a very low risk of serious complications. Following complications rates have been reported after TVT: bladder perforation 3,8%, urinary tract infection 4,1%, complications requiring laparotomy 3,4%, complete postoperative urinary retention 2,3% and minor voiding difficulties 7,6%. All these complications or side effects occur in up to 20 - 30% of the patients. Long-term effects of TVT are still unclear and complications such as vaginal erosion or urinary tract protrusion of the tape are concerning.

   Bulking agents create an artificial mass into the urethral submucosa and according to hypothesis improve urethral coaptation and restore continence especially when abdominal pressure is increased. It has also been suggested that midurethral injection therapy may increase the central filler volume and consequently increase the power of the urethral sphincter. Several different agents have been used for periurethral and transurethral injections, e.g. collagen, ethylene vinyl alcohol, hyaluronic acid and polyacrylamide hydrogel (PAHG). However, some of these agents have been abandoned due to safety issues.

   In Nordic countries Polyacrylamide hydrogel (PAHG) is nowadays used for urethral injections. PAHG is biocompatible, non-biodegradable, non-allergenic, non-migrational, atoxic, stable, and sterile. Urethral bulking therapy is minimally invasive in nature and treatment doesn't require hospitalization. Procedure can be performed under local anaesthesia.

   The efficacy of PAHG-injections in treating stress urinary incontinence has varied from 64% to 74% depending on the treated patient group. Urethral injections have a lower risk of complications than TVT-operation and PAHG has shown a very low risk of serious adverse events. Bulking therapy has no negative effect in terms of possible subsequent midurethral sling operation.

   Cochrane review on urethral injection therapies concluded that injection therapies are inferior to surgery at 1-year follow-up but have a better safety profile. However, the objective outcome and effect of the treatment are not necessarily equal to patient satisfaction and improvement in quality of life (QOL). A study by Corcos et al. comparing surgery and collagen injections for treatment of SUI showed significantly better outcome in 24-hour pad test for women treated with surgery compared to those treated with collagen injections but no difference in patient satisfaction and QOL at 12 months between the two groups. Number and severity of complications were much greater in the surgery group. A questionnaire study assessing treatment acceptability and treatment expectations in women with lower urinary tract symptoms, showed that patients have a general preference for less invasive therapy even with the cost of lower success rate.
2. Hypothesis and aims of the study

   Randomized studies comparing urethral injection treatment and TVT are missing. There was no significant difference in patient satisfaction after urethral injections with collagen and surgery. Surgical group in this study consisted of treatment with sling operation, Burch procedure or needle bladder neck suspensions. While there are no comparative studies between TVT and Bulkamid®, the knowledge about cost-effectiveness and patient satisfaction is missing.

   This prospective randomized study compares TVT and Bulkamid®-injections in treatment of SUI.
3. Materials and methods

Subjects included in this study are women suffering from such a stress urinary incontinence that a non-conservative treatment is planned. They have to be willing to participate in the study.

Patients are given oral and written information on the study and randomized into two groups undergoing either TVT-Exact® or Bulkamid®.

Study Flow:

1. Randomization before treatment
2. Treatment (Bulkamid or TVT exact)
3. Phone call contact after 1 month
4. Second Bulkamid-treatment if necessary within 3 months after first treatment
5. 3 months follow-up visit and decisions about secondary treatment if necessary
6. (Secondary) TVT treatment at least 3 months after follow-up visit (or Bulkamid treatment following primary TVT-treatment)
7. One-year follow-up visit and decisions about further treatments if necessary (re-Bulkamid/TVT?)
8. Questionnaires 2,3 and 4-years after treatment, mail contact
9. 3-year follow-up visit offered
10. 5-year follow-up visit

Examinations before treatment:

* 2-3 day micturition diary and standardised questionnaire forms assessing symptom distress (UDI-6, IIQ-7) and the impact of urinary incontinence on quality of life and sexual function (RAND-36, PISQ-12)
* Patient's estimation of the distress caused by SUI (VAS scale 0= no distress to 10= very much distress)
* Exclusion of urinary tract infection (sample 2-3 weeks before treatment)
* Physical examination: cough stress test and PVR measurement by ultrasound, exclusion of pelvic organ prolapse and large uterine myomas
* Urodynamics, if needed to confirm diagnosis
* A stress pad test described by Svenningsen et al.20 (Pad weighing after 20 jumping jacks on the spot and three forceful coughs in the standing position with 300 ml bladder volume. To women unable to perform the test it was modified version to 10 coughs in the standing position).

Examinations after the treatment:

* Post-void residual urine volume (if <150ml patient will be discharged)
* Pain in VAS scale (0=no pain to 10= worst possible pain the patient can imagine)
* Question of: would the patient recommend the treatment to a good friend?
* Was the pain during treatment: as the patient expected, less, worse?

Examinations on follow-up visits (3 months, 1 year, 3 years, 5 years):

* Gynecological examination (with ultrasound)
* Cough stress test with 200 to 250 filling in the bladder
* Stress PAD test described earlier
* PVR measurement
* Exclusion of urinary tract treatment to patients with failed response or symptoms of infection
* Questionnaires (RAND-36, UDI 6, IIQ-7)
* Pain in VAS scale
* Satisfaction to treatment in VAS scale
* Question of: would the patient recommend the treatment to a good friend?
* The length of sick-leave after the operation, possible other visit to other health care providers
* Analysis of the efficacy of the treatment against stress urinary incontinence in categories: fully recovered, partly recovered, no change, worse symptoms, cannot answer.

The surgeon, who performed the procedure, will not perform follow-up visits.Questionnaires (RAND 36, UDI-6, IIQ-7, PISQ-12) will be collected from the patients two to four years after treatment via mail. Also above mentioned analysis of the efficacy of the treatment and further questions on possible incontinence are collected.

The analysis of possible adverse events (complications) of the treatment will be performed during the operation and after it during the whole follow-up time. The adverse effects will be categorized as related to the treatment, possibly related to the treatment and not related to the treatment.

TVT treatment

TVT will be performed under local anesthesia (70 - 100 ml 0.25% prilocain cum epinephrine) with i.v. pain medication phentanyl two doses and more on request. Operation will be performed with TVT-Exact® kit. Operation can be performed policlinically or in an operation theatre depending on the patient's medical condition. Cystoscopy will be performed after the set of tapes. A cough stress test with 250 to 300 ml bladder fulfillment will show the right tension of the tape. Before the operation a prophylactic antibiotic of Cefuroxime 1.5 g i.v will be given (Dalacin 900 mg i.v in cases of allergy to penicillin). The patient can go home after 2 to 4 hours follow-up, when PVR is under 150 ml. A sick leave of 5 days is recommended.

All used medications, the duration of treatment, follow-up time and the time when patients leave the hospital are written down as well as the onset of urination. Pain is asked in VAS scale 0 to 10 (maximal and total VAS) and the patient's are asked to describe, whether the pain during treatment was as expected/less/more.

Bulkamid®- injections

Urethral injections will be performed policlinically under local anesthesia (10 ml lidocain, two injections on both sides of the urethra). The Bulkamid-injections will be transurethral four injections (0.2 - 1ml) in locations "ten, two and five and seven o'clock" within 0.5 to 1 cm from the bladder - urethra junction.

Additional injections will be avoided and can be injected only if the first injections fail. After the operation the patient urinates to empty the bladder. The PVR is checked after the treatment with ultrasound simultaneously with evaluation of stability of the Bulkamid-injections. The treatment will be photographed as before and after still pictures for later evaluation.

All used medications, the duration of treatment, follow-up time and the time when patients leave the hospital are written down as well as the onset of urination. Pain is asked in VAS scale 0 to 10 (maximal and total VAS) and the patient's are asked to describe, whether the pain during treatment was as expected/less/more.

If the given treatment fails to treat stress urinary incontinence or stress urinary incontinence returns after a while, a TVT- or Bulkamid®-operation can be (re-)performed after the follow-up visit. The primary treatment after one Bulkamid®-injection is a secondary injection after follow-up visit. Bulkamid® injections do not interfere subsequent TVT operation and vice versa.

Re-injections of Bulkamid will be done in basis of "filling up the gaps" after primary treatment. In other words they are done according to the situation seen during second treatment. The treatments are photographed before and after (still pictures).

Sample size

The study will be conducted as a non-inferiority trial based on patient satisfaction rates. The patient satisfaction rate of VAS scale ≥80 was assumed in 80% and 75% of the TVT- and Bulkamid-patients. If there is a true difference in favour of the standard treatment of 5%, then 192 patients (96 per group) are required to be 80% sure that the upper limit of a one-sided 95% confidence interval will exclude a difference in favour of the standard group of more than 20%. A 10% dropout rate was assumed and 212 women were planned to randomize (1:1) in this study.

Randomization numbers

The randomization numbers will be generated before the onset of the study and sealed in opaque envelopes. Randomization will performed using a computer-assisted random block system (R Development Core Team, 2006, Greg Snow, 2006) with permuted randomization for random block clinical trials. Random blocks of 4 to 6 women were used. Altogether 250 random numbers will be generated.

Time schedule

The enrollment of the patients will be done within the end of year 2017. Primary follow-up and reporting of first outcomes will happen within 2018.

Ethical reason

The effectiveness or complications of operations for stress urinary incontinence have been shown, but a randomized comparison of TVT and urethral injection is missing. Therefore this study is needed. This study will also provide information about the cost-effectiveness and patient satisfaction of these treatments. This is a comparison between a more effective TVT operation that has a higher risk for complications and a probably less effective, but safer Bulkamid®- injections. TVT operation can be performed after Bulkamid® treatment and Bulkamid® injections do not interfere the subsequent TVT treatment.

ELIGIBILITY:
Inclusion Criteria:

* No previous stress urinary incontinence operation
* Positive cough stress test without urge-type urine leakage
* Post-void residual urine volume (PVR) <100ml
* Urine bladder capacity >3dl in 3-day micturition diary.

Exclusion Criteria:

* BMI >35 kg/m2
* Neurogenic disease which can be associated with bladder disorders
* Use of anticholinergics or mirabegrone
* Illness or condition causing even a relative risk for complications in TVT operation (e.g. lower urinary tract anomaly, previous radiation therapy of the pelvis, anticoagulation or haemophilia)
* Active malignancy
* Current UTI or recurrent UTI (over 3 episodes within the past year)
* Urogenital prolapse of more than second degree
* Pregnancy or future plans of pregnancy
* Inability to understand purpose of the study
* Uterine myoma requiring operational treatment
* Autoimmune or connective tissue disease contraindicating operation

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction to treatment | Up to 5 years after treatment
  Patient satisfaction measured on VAS scale of 0 (extremely unsatisfied) to 100 (extremely satisfied). VAS ≥80 was defined as a good level of satisfaction. Patient satisfaction is measured on follow-up visits (3 months, 1 year, 3 years, 5 years).
Complications of the treatment | Up to 5 years after treatment
  Possible complications are listed after treatment and on follow-up visits.
Effectiveness of the treatment in reducing urinary leakage | Up to 5 years after treatment
  A stress pad test (Pad weighing after 20 jumping jacks on the spot and three forceful coughs in the standing position with 300 ml bladder volume. To women unable to perform the test it was modified version to 10 coughs in the standing position) performed before treatment and on follow-up visits (3 months, 1 year, 3 years, 5 years).

SECONDARY OUTCOMES:
Cost-effectiveness of the treatment | Up to 5 years after treatment
  Questionnaires including UDI-6, IIQ-7,RAND-36, PISQ-12
Pain during and after treatment | Up to 5 years after treatment
  VAS scale 0-10 used.
Changes in Quality of Life and symptoms | Up to 5 years after treatment
  Questionnaires including UDI-6, IIQ-7,RAND-36, PISQ-12

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki Women's Hospital, Helsinki, Finland

REFERENCES:
- [Background] Bezerra CA, Bruschini H, Cody DJ. Traditional suburethral sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD001754. doi: 10.1002/14651858.CD001754.pub2. PMID 16034866
- [Background] Rehman H, Bezerra CC, Bruschini H, Cody JD. Traditional suburethral sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD001754. doi: 10.1002/14651858.CD001754.pub3. PMID 21249648
- [Background] Nilsson CG, Palva K, Aarnio R, Morcos E, Falconer C. Seventeen years' follow-up of the tension-free vaginal tape procedure for female stress urinary incontinence. Int Urogynecol J. 2013 Aug;24(8):1265-9. doi: 10.1007/s00192-013-2090-2. Epub 2013 Apr 6. PMID 23563892
- [Background] Laurikainen E, Valpas A, Aukee P, Kivela A, Rinne K, Takala T, Nilsson CG. Five-year results of a randomized trial comparing retropubic and transobturator midurethral slings for stress incontinence. Eur Urol. 2014 Jun;65(6):1109-14. doi: 10.1016/j.eururo.2014.01.031. Epub 2014 Jan 31. PMID 24508070
- [Background] Kuuva N, Nilsson CG. A nationwide analysis of complications associated with the tension-free vaginal tape (TVT) procedure. Acta Obstet Gynecol Scand. 2002 Jan;81(1):72-7. doi: 10.1034/j.1600-0412.2002.810113.x. PMID 11942891
- [Background] Abbott S, Unger CA, Evans JM, Jallad K, Mishra K, Karram MM, Iglesia CB, Rardin CR, Barber MD. Evaluation and management of complications from synthetic mesh after pelvic reconstructive surgery: a multicenter study. Am J Obstet Gynecol. 2014 Feb;210(2):163.e1-8. doi: 10.1016/j.ajog.2013.10.012. Epub 2013 Oct 11. PMID 24126300
- [Background] Kerr LA. Bulking agents in the treatment of stress urinary incontinence: history, outcomes, patient populations, and reimbursement profile. Rev Urol. 2005;7 Suppl 1(Suppl 1):S3-S11. PMID 16985874
- [Background] Kuhn A, Stadlmayr W, Lengsfeld D, Mueller MD. Where should bulking agents for female urodynamic stress incontinence be injected? Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jun;19(6):817-21. doi: 10.1007/s00192-007-0535-1. PMID 18157642
- [Background] Klarskov N, Lose G. Urethral injection therapy: what is the mechanism of action? Neurourol Urodyn. 2008;27(8):789-92. doi: 10.1002/nau.20602. PMID 18642372
- [Background] Kirchin V, Page T, Keegan PE, Atiemo K, Cody JD, McClinton S. Urethral injection therapy for urinary incontinence in women. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD003881. doi: 10.1002/14651858.CD003881.pub3. PMID 22336797
- [Background] Lose G, Sorensen HC, Axelsen SM, Falconer C, Lobodasch K, Safwat T. An open multicenter study of polyacrylamide hydrogel (Bulkamid(R)) for female stress and mixed urinary incontinence. Int Urogynecol J. 2010 Dec;21(12):1471-7. doi: 10.1007/s00192-010-1214-1. Epub 2010 Jul 20. PMID 20645077
- [Background] Leone Roberti Maggiore U, Alessandri F, Medica M, Gabelli M, Venturini PL, Ferrero S. Outpatient periurethral injections of polyacrylamide hydrogel for the treatment of female stress urinary incontinence: effectiveness and safety. Arch Gynecol Obstet. 2013 Jul;288(1):131-7. doi: 10.1007/s00404-013-2718-y. Epub 2013 Feb 1. PMID 23371485
- [Background] Toozs-Hobson P, Al-Singary W, Fynes M, Tegerstedt G, Lose G. Two-year follow-up of an open-label multicenter study of polyacrylamide hydrogel (Bulkamid(R)) for female stress and stress-predominant mixed incontinence. Int Urogynecol J. 2012 Oct;23(10):1373-8. doi: 10.1007/s00192-012-1761-8. Epub 2012 Apr 25. PMID 22531952
- [Background] Sokol ER, Karram MM, Dmochowski R. Efficacy and safety of polyacrylamide hydrogel for the treatment of female stress incontinence: a randomized, prospective, multicenter North American study. J Urol. 2014 Sep;192(3):843-9. doi: 10.1016/j.juro.2014.03.109. Epub 2014 Apr 2. PMID 24704117
- [Background] Mouritsen L, Lose G, Moller-Bek K. Long-term follow-up after urethral injection with polyacrylamide hydrogel for female stress incontinence. Acta Obstet Gynecol Scand. 2014 Feb;93(2):209-12. doi: 10.1111/aogs.12283. Epub 2013 Dec 24. PMID 24372312
- [Background] Koski ME, Enemchukwu EA, Padmanabhan P, Kaufman MR, Scarpero HM, Dmochowski RR. Safety and efficacy of sling for persistent stress urinary incontinence after bulking injection. Urology. 2011 May;77(5):1076-80. doi: 10.1016/j.urology.2010.10.010. Epub 2011 Jan 8. PMID 21216448
- [Background] Corcos J, Collet JP, Shapiro S, Herschorn S, Radomski SB, Schick E, Gajewski JB, Benedetti A, MacRamallah E, Hyams B. Multicenter randomized clinical trial comparing surgery and collagen injections for treatment of female stress urinary incontinence. Urology. 2005 May;65(5):898-904. doi: 10.1016/j.urology.2004.11.054. PMID 15882720
- [Background] Svenningsen R, Staff AC, Schiotz HA, Western K, Kulseng-Hanssen S. Long-term follow-up of the retropubic tension-free vaginal tape procedure. Int Urogynecol J. 2013 Aug;24(8):1271-8. doi: 10.1007/s00192-013-2058-2. Epub 2013 Feb 16. PMID 23417313
- [Derived] Freitas AI, Isaksson C, Rahkola-Soisalo P, Mentula M, Mikkola TS. Tension-Free Vaginal Tape versus Polyacrylamide Hydrogel Injection for Stress Urinary Incontinence - 5-Year Follow-Up. NEJM Evid. 2025 May;4(5):EVIDoa2400216. doi: 10.1056/EVIDoa2400216. Epub 2025 Apr 22. PMID 40261117
- [Derived] Itkonen Freitas AM, Isaksson C, Rahkola-Soisalo P, Tulokas S, Mentula M, Mikkola TS. Tension-Free Vaginal Tape and Polyacrylamide Hydrogel Injection for Primary Stress Urinary Incontinence: 3-Year Followup from a Randomized Clinical Trial. J Urol. 2022 Sep;208(3):658-667. doi: 10.1097/JU.0000000000002720. Epub 2022 Aug 5. PMID 35942796